CLINICAL TRIAL: NCT04967079
Title: Combined MEK Inhibitor Trametinib and RTK Inhibitor Anlotinib Therapy in Non-G12C KRAS-Mutant Non-Small Cell Lung Cancer Patients
Brief Title: Trametinib Plus Anlotinib in Non-G12C KRAS-Mutant NSCLC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Director of department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATRAS-LC
Record Dates: First submitted 2021-07-05; First posted 2021-07-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non-G12C KRAS Mutations; Advanced NSCLC; MEK inhibitor-trametinib; RTKs inhibitor-Anlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trametinib; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trametinib + Anlotinib (Experimental): Anlotinib given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) plus trametinib 2 milligrams (mg) given orally, once daily.
  Interventions: Drug: Trametinib; Drug: Anlotinib

INTERVENTIONS:
Drug: Trametinib — Trametinib 2 mg given orally, once daily
Drug: Anlotinib — Anlotinib given orally, every two weeks followed by a one-week discontinuation cycle

SUMMARY:
This is a Phase I exploratory study. The study is divided into two parts (A/B).In part A, the primary endpoint is the determination of the recommended phase 2 dose (RP2D). Secondary endpoint for phase Ia includes evaluating the objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and adverse events (AEs). Following the establishment of the RP2D, the expansion cohort will be initiated.

Transitioning to part B, 20 patients will be enrolled to further evaluate the ORR. All patients will receive the trametinib plus anlotinib regimen based on the RP2D determined in part A. The primary endpoint for part B is to assess the ORR, while secondary endpoint includes evaluating PFS, overall survival (OS), DCR, AEs, and duration of overall response (DoR).

In part A, the study plans to enroll eligible patients to receive the MEK inhibitor trametinib (2 mg) in combination with anlotinib (6mg, 8 mg, 10 mg, 12 mg). The number of subjects is determined according to the actual situation of dose climbing.

In part B, another 20 eligible patients will be enrolled and treated with trametinib (2mg) + anlotinib (RP2D), until the disease progression (PD) or unacceptable toxicity occurs to further evaluate the safety, tolerability and efficacy.

Patients participated in safety follow-up after the first course of treatment until 3 months after discontinuation due to PD or toxicity. Dose-limiting toxicities from the first cycle were collected. Therapeutic efficacy evaluation was scheduled according to RECIST version 1.1 every 4-8 weeks. After the investigators' evaluation, the assessment cycle could extend to 12 weeks or longer due to the uncontrollable factors during the treatment period. Blood samples will be collected for pharmacokinetic analysis and biomarker discovery at baseline and at each periodic assessment.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study subjects should fulfill the following criteria:

  1. According to the 8th edition of the American Journal of Critical Care (AJCC)/Union for International Cancer Control (UICC) Tumor Node Metastasis (TNM) NSCLC staging system, locally advanced (stage III B/III C), metastatic or recurrent (stage IV) NSCLC patients confirmed by histology or cytology. The NSCLC patient cannot receive surgery and radical radiotherapy, and at least one measurable lesion is confirmed according to RECIST 1.1.
  2. KRAS mutation positive excluded KRASG12C mutation.
  3. No active brain metastases.
  4. Age ≥18 years old and ≤75 years old.
  5. ECOG PS score: 0-1.
  6. Patients who had previously received at least 1st-line standard therapy. Note: the treatment naïve patients who refused immunotherapy/chemotherapy at 1st-line, and willingly enrolled in the clinical trial are also eligible.

     Part A: advanced NSCLC patients with non-G12C mutations who have previously received standard treatment or treatment naïve. Part B: advanced NSCLC patients with non-G12C mutations who have previously received standard 1st or more treatment.
  7. Palliative radiotherapy must be completed 7 days before the first dose of study drug is administered.
  8. The main organs are functioning normally, that is, they meet the following standards:

     Good hematopoietic function, defined as absolute neutrophil count ≥1.5 billion

     /L, platelet count ≥100 billion/L, hemoglobin ≥90 g/L [no blood transfusion or no erythropoietin (EPO) within 7 days before enrollment dependence]; The biochemical test results should meet the following standards: BIL <1.25 times the upper limit of normal (ULN); ALT and AST <2.5×ULN; if liver metastasis occurs, ALT and AST <5×ULN; Cr ≤1.5×ULN or creatinine clearance Rate (CCr) ≥60 ml/min; good coagulation function, International Normalized Ratio (INR) and PT ≤1.5 times of ULN; if the subject is receiving anticoagulation therapy, PT should be within the prescribed range of anticoagulation drugs; Women of childbearing age should agree to take contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study and within 6 months after the study; the serum or urine pregnancy test of non-breastfeeding patients should be negative; male patients should agree to take contraceptive measures during the study period and within 6 months after the study.
  9. The patients voluntarily participated in the study, signed an informed consent form and had good compliance.
  10. The expected survive time is longer than 3 months.

Exclusion Criteria:

* Subjects must not enter the study if any of the following exclusion criteria are fulfilled:

  1. Patients with active central nervous system metastasis are excluded. If a subject has received adequate treatment for central nervous system (CNS) metastasis at least 2 weeks before enrollment, and is neurologically restored to baseline levels (except for residual signs or symptoms related to CNS treatment), the subject is eligible. In addition, subjects must stop corticosteroids, or the daily dose of prednisone must be stabilized orgradually reduced to ≤10 mg (or equivalent dose).
  2. Small cell lung cancer (including mixed small cell and non-small cell lung cancer) or hollow central squamous cell carcinoma.
  3. There are obvious bleeding symptoms.
  4. Patients who have previously received MEK inhibitors, anlotinib or other multi-targeted anti-angiogenic therapy.
  5. Patients with dysphagia, gastrointestinal resection, chronic diarrhea, intestinal obstruction and other factors that affect oral medication.
  6. Patients who are known to have active brain metastases, spinal cord compression, cancerous meningitis, brain or soft tissue diseases diagnosed by computed tomography (CT) or magnetic resonance imaging (MRI) at the time of screening.
  7. Patients with severe and/or uncontrollable diseases, such as: unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months, severe uncontrollable arrhythmia; uncontrolled blood pressure (BP, constriction BP > 140 mmHg, diastolic BP > 90 mmHg).
  8. Active or uncontrolled serious infections.
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis.
  10. Incomplete control of eye inflammation or eye infection, or any condition that may cause the above eye diseases.
  11. Poor diabetes control (fasting blood glucose (FBG) > 10 mmol/L).
  12. Routine urine test results show that urine protein is ≥++, and the 24-hour urine protein quantitative is> 1.0 g.
  13. Active tuberculosis.
  14. Uncontrollable hypercalcemia (calcium ion> 1.5 mmol/L or calcium> 12 mg/dL or corrected serum calcium >ULN), or symptomatic hypercalcemia that requires continued bisphosphonate therapy.
  15. Long-term unhealed wounds or fractures.
  16. Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders.
  17. Patients with known severe allergies (≥Grade 3) to active ingredients and excipients.
  18. Patients who also suffer from other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.); patients who have been assessed by the investigator as having concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.
  19. During the clinical trial, the subjects or their sexual partners cannot or refuse to take effective contraceptive measures.
  20. Pregnant or breastfeeding women.
  21. Previous treatment including Chinese medicine treatment.
  22. Patients who are allergic to any medicine or any ingredient.
  23. In other cases, patients who are not eligible for inclusion as assessed by the investigator.
  24. The expected survive time is shorter than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Part A: Recommended phase 2 dose (RP2D) | 1 year
  The determination of RP2D relied on several priority indexes: firstly, the MTD, followed by ORR, and mean tumor shrinkage rate. If the highest dose of anlotinib (12 mg) did not reach MTD, ORR would be the main index for defining the RP2D. Subsequently, if 2 or more dosage groups had same ORR, the average tumor shrinkage rate would replace MTD and ORR in determining RP2D.
Part B: Objective response rate (ORR) | 1.5 year
  Percentage of participants achieving CR and PR.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  The time from the start of systemic treatment date to the date of first documented disease progression (event: disease progression - DP, based on RECIST, death, adverse events, which provide to disqualification from further therapy).
Disease control rate (DCR) | 2 years
  Percentage of participants achieving CR and PR and SD.
Overall survival (OS) | 2 years
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Adverse Event (AE) | 2 years
  Adverse event caused by the combination treatments.
Duration of overall response (DoR) | 2 years
  The time from date of the first documentation of objective response (CR or PR) to the first documentation of PD or to death due to any cause in the absence of documented PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No